CLINICAL TRIAL: NCT05345535
Title: Investigation of the Acute Effects of Trampoline Exercises on Balance, Proprioception, Vertical Jump and Cognitive Functions
Brief Title: Acute Effects of Trampoline Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Elif Dinler, Research Assistant, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/033
Record Dates: First submitted 2022-04-19; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Exercise; Aerobic Exercise
Keywords: Balance; Joint position sense; Myoton; Foot and ankle
MeSH Terms: conditions — Motor Activity | interventions — Walking

STUDY DESIGN:
Intervention Model Description: Two randomized controlled group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants of study group will perform 45 minutes of trampoline exercises. Evaluations are going to be done immediately before and after trampoline session.
  Interventions: Other: Trampoline exercise
- Control group (Experimental): Participants of control group will perform 45 minutes of walking. Evaluations are going to be done immediately before and after walking session.
  Interventions: Other: Walking

INTERVENTIONS:
Other: Trampoline exercise — 45 minutes of exercises that includes upper and lower extremity movements a trampoline with music
  Arms: Study group
Other: Walking — 45 minutes of moderate tempo walking
  Arms: Control group

SUMMARY:
The aim of the study is to investigate the acute effects of trampoline exercises on balance, proprioception, vertical jump and cognitive functions. As a result of the study, it is thought that trampoline exercises will affect balance, proprioception, vertical jump, cognitive functions and myotonometric properties of the muscle more positively than walking.

DETAILED DESCRIPTION:
30 healthy, volunteer women who meet the inclusion criteria will be included in the study. Participants will be divided into two group randomly. The women in the study group will be evaluated before the first trampoline exercise sessions and the acute effect will be evaluated by re-evaluating at the end of the 45-minute (min) session. The control group women will be evaluated and after 45 minutes of walking, they will be evaluated again for the acute effect over the relevant parameters. The evaluations to be made to the participants are given below;

* Demographic Information Form (Age, height (cm), weight (kg), occupation, education level, previous and present diseases, smoking, etc.)
* Balance Evaluation - Y Balance Test
* Ankle joint position sense - Electrogoniometer
* Cognitive assessment - Stroop test
* Vertical jump test - tape measure
* Myotonometric properties of gastrocnemius, tibialis anterior and peroneal muscles- Myoton device

ELIGIBILITY:
Inclusion Criteria:

* Females who agreed to participate in the study voluntarily,
* Female individuals between the ages of 18-65 years old
* Females who have mini mental test score more than 25

Exclusion Criteria:

* Those with a Body Mass Index (BMI) greater than 30 kg/m²,
* Pregnant women,
* Those with following problems; neural findings, malignancy, inflammation, arthritis, metabolic bone disease, column vertebralis or lower extremity surgery, cardiovascular system diseases, severe osteoporosis, communication and hearing disorders, chronic diseases such as diabetes, hypertension,
* Those who illiterate,
* Individuals who do sports for more than 150 minutes a week,
* Individuals with a professional sports background, Individuals who do sports for more than 150 minutes a week
* Individuals with a professional sports background

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Y balance test score | Immediately after the intervention
  Balance score is going to be assess by Y balance test to determine change from baseline.
Change from baseline in ankle position sense degree | Immediately after the intervention
  Ankle position sense degree is going to be assess by electroconiometer to determine change from baseline.
Change from baseline in vertical jump distance | Immediately after the intervention
  Vertical jump distance (centimeter) is going to be assess by vertical jump test by a tape measure.
Change from baseline in myotonometric characteristics | Immediately after the intervention
  Myotonometric characteristic is going to be assess by MyotonPRO device.

SECONDARY OUTCOMES:
Change from baseline in cognitive status | Immediately after the intervention
  Cognitive status is going to be assess by Stroop Test. Correct and false answers will be record. More correct answer shows higher cognitive status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No